CLINICAL TRIAL: NCT04980222
Title: A Phase II Study Evaluating the Safety and Efficacy of Glofitamab in Combination With Rituximab (R) Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP) in Circulating Tumor (ct)DNA High-Risk Patients With Untreated Diffuse Large B-Cell Lymphoma
Brief Title: A Study to Evaluate the Safety and Efficacy of Glofitamab in Combination With Rituximab (R) Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP) in Circulating Tumor (ct)DNA High-Risk Patients With Untreated Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO43075; 2023-504994-19-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — glofitamab; tocilizumab; Doxorubicin; Vincristine; Prednisone; Rituximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Glofitamab + R-CHOP Immunochemotherapy (Experimental): Participants will receive step-up doses of glofitamab, starting on Day 8 of Cycle 3 (2.5 mg), Day 15 of Cycle 3 (10 mg), then 30 mg glofitamab will be given every three weeks (Q3W) onwards, on Day 8 of Cycles 4-6 and on Day 1 of Cycles 7-10. (cycle length = 21 days)
  Participants will receive rituximab, cyclophosphamide, doxorubicin, and vincristine Q3W on Day 1 of Cycles 1-6. Prednisone or prednisolone will be administered daily (QD) on Days 1-5 of Cycles 1-6. (cycle length = 21 days)
  Interventions: Drug: Glofitamab; Drug: Tocilizumab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Rituximab; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Glofitamab — Participants will receive intravenous (IV) glofitamab as per schedule specified in the treatment arm.
Drug: Tocilizumab — Participants will receive tocilizumab as needed to manage cytokine release syndrome (CRS).
Drug: Doxorubicin — Participants will receive 50 mg/m2 body surface area of doxorubicin IV as per schedule specified in the treatment arm.
Drug: Vincristine — Participants will receive 1.4 mg/m2 body surface area of vincristine IV as per schedule specified in the treatment arm.
Drug: Prednisone — Participants will receive 100 mg of prednisone or prednisolone as per schedule specified in the treatment arm.
Drug: Rituximab — Participants will receive 375 mg/m2 body surface area of rituximab IV as per schedule specified in the treatment arm.
Drug: Cyclophosphamide — Participants will receive 750 mg/m2 body surface area of cyclophosphamide IV as per schedule specified in the treatment arm.

SUMMARY:
This Phase II, open-label, multicenter study will evaluate the safety, efficacy, and pharmacokinetics of glofitamab in combination with rituximab in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in individuals with circulating tumor DNA (ctDNA) high-risk diffuse large B-cell lymphoma (DLBCL), as the first line of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with CD20-positive DLBCL, including one of the following diagnoses made according to the 2016 World Health Organization (WHO) classification of lymphoid neoplasms

  * DLBCL, not otherwise specified, including GCB and ABC/non-GCB types as well as double-expressor lymphoma (coexpression of MYC and BCL2)
  * High-grade B-cell lymphoma (HGBCL) with MYC and BCL2 and/or BCL6 translocations
  * Patients with de novo transformed follicular lymphoma (patients with discordant bone marrow involvement, i.e., evidence of low-grade histology in bone marrow) may be considered after discussion with the Medical Monitor
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* International Prognostic Index (IPI): 2-5
* Life expectancy of at least 6 months
* Adequate biomarker blood samples prior to initiation of R-CHOP on Day 1 of Cycle 1 and on Day 1 of Cycle 2 submitted for screening for determination of ctDNA status
* At least one bi-dimensionally fluorodeoxyglucose (FDG)-avid measurable lymphoma lesion on positron emission tomography/computed tomography (PET/CT) scan
* Left ventricular ejection fraction (LVEF) >=50%, as determined on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Adequate hematopoietic function
* Contraception use

Additional Inclusion Criterion for ctDNA High-Risk Participants:

* Plasma sample evaluated to be ctDNA high risk

Exclusion Criteria:

* Current diagnosis of B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classic Hodgkin lymphoma (gray-zone lymphoma), primary mediastinal (thymic) large B-cell lymphoma, T-cell/histiocyte-rich large B-cell lymphoma, Burkitt lymphoma, central nervous system (CNS) lymphoma (primary or secondary involvement), primary effusion DLBCL, and primary cutaneous DLBCL
* Contraindication to any of the individual components of R-CHOP, including prior receipt of anthracyclines, history of severe allergic or anaphylactic reactions to murine monoclonal antibodies, or known sensitivity or allergy to murine products
* Prior treatment for indolent lymphoma
* Prior solid organ or allogeneic stem cell transplant
* Prior therapy for DLBCL and high-grade B-cell lymphoma (HGBCL) with the exception of palliative, short-term treatment with corticosteroids
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 12 months after the final dose of R-CHOP, 3 months after the final dose of tocilizumab (if applicable), or 2 months after the final dose of glofitamab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
End of Treatment Complete Response (EOT CR) Rate | Up to approximately 24 months

SECONDARY OUTCOMES:
Overall Response Rate (ORR) at the EOT | Up to approximately 24 months
Progression-free Survival (PFS) | Up to approximately 24 months
Overall Survival (OS) | Up to approximately 24 months
Percentage of Participants with Adverse Events (AEs) | Up to 90 days after the final dose of study treatment
Serum Concentration of Glofitamab | At pre-defined intervals up to approximately 10 months
Maximum Concentration (Cmax) of Glofitamab | At pre-defined intervals up to approximately 10 months
Total Exposure (AUC) of Glofitamab | At pre-defined intervals up to approximately 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- United States (8):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - University of Iowa, Iowa City, Iowa
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Baylor University Medical Center, Dallas, Texas
- Aarhus Universitetshospital Skejby, Aarhus N, Denmark
- France (2):
  - Hopital Henri Mondor, Créteil
  - Centre Henri Becquerel, Rouen
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk
  - Uniwersytecki Szpital Kliniczny; Klinika Hematologii, Nowotworów Krwi i Transplantacji Szpiku, Wroclaw
- Spain (4):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing